CLINICAL TRIAL: NCT05851911
Title: Children's Hospital of Chongqing Medical University
Brief Title: Passive Transmission of COVID-19 Antibody From Mother to Infant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, yuting yang, researcher, Children's Hospital of Chongqing Medical University
Other Study IDs: 2022-380
Record Dates: First submitted 2023-05-09; First posted 2023-05-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Passive Transmission of Maternal and Infant Antibodies
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group 1: Mother not vaccinated with COVID-19 vaccine
  Interventions: Biological: sars-cov-2 vaccine or infection
- Control group 2: The mother was vaccinated with COVID-19 vaccine before pregnancy, and was not infected during pregnancy
  Interventions: Biological: sars-cov-2 vaccine or infection
- Control group 3: The mother was vaccinated with COVID-19 vaccine before pregnancy, and was infected during pregnancy
  Interventions: Biological: sars-cov-2 vaccine or infection
- Experimental group: The mother was not vaccinated with COVID-19 vaccine before pregnancy, so she was infected during pregnancy
  Interventions: Biological: sars-cov-2 vaccine or infection

INTERVENTIONS:
Biological: sars-cov-2 vaccine or infection — Whether to vaccinate COVID-19 vaccine, or infect with sars-cov-2

SUMMARY:
At present, there is no relevant research focusing on children's acquisition of novel coronavirus antibodies through maternal passive transmission. Therefore, this study assessed the changes of maternal passive transmission of COVID-19 antibodies by monitoring the specific antibodies of COVID-19 in young children; This will lay a foundation for further exploring the risk of COVID-19 infection in children and formulating immune prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0-2;
2. No history of blood transfusion, chemotherapy, or related immunosuppressive therapy; No immune system related diseases;

Exclusion Criteria:

Not willing to participate

Ages: 0 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Samples of infants not infected with COVID-19 and not vaccinated with COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 IgG | duration of time over which each participant could be 6-month to 12-month
  ELISA detection of SARS-CoV-2 IgG antibody levels
SARS-CoV-2 neutralizing antibody | duration of time over which each participant could be 6-month to 12-month
  detection the level of SARS-CoV-2 neutralizing antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Yuting Yang, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Contact the project leader